CLINICAL TRIAL: NCT00013806
Title: CHP677: I-Metaiodobenzylguanidine (I-MIBG) Therapy for Refractory Neuroblastoma: a Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Purpose: Treatment
Other Study IDs: NCRR-M01RR00240-1748
Record Dates: First submitted 2001-03-29; First posted 2001-03-30 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Neuroblastoma
Keywords: Relapsed and refractory neuroblastoma
MeSH Terms: conditions — Neuroblastoma; Recurrence | interventions — 3-Iodobenzylguanidine

INTERVENTIONS:
Drug: 131I-MIBG

SUMMARY:
131I-metaiodobenzylguanidine (131I-MIBG) is a norepinephrine analog that concentrates in adrenergic tissue and therefore holds promise for cell-specific treatment of neuroblastoma. This is a dual institution, Phase II study of 131I-MIBG administered at the previously defined maximum practical dose of 18 mCi/kg to children with relapsed or refractory neuroblastoma.

ELIGIBILITY:
Inclusion criteria: Refractory neuroblastoma with original diagnosis based on tumor histopathology or elevated urine VMA with typical tumor cells in the bone marrow.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States